CLINICAL TRIAL: NCT04023747
Title: Oxford Pre-cancerous Lymphoproliferative Disorders: Analysis and Interception Study
Brief Title: Oxford Pre-cancerous Lymphoproliferative Disorders Study
Acronym: OxPLoreD
Status: Active, not recruiting | Type: Observational
Sponsor: University of Oxford (Other)
Collaborators: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: OCTO_091
Record Dates: First submitted 2019-06-25; First posted 2019-07-17 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2024-10

CONDITIONS: Pre-cancerous Lymphoproliferative Disorders
Keywords: Monoclonal B-Cell Lymphocytosis; Asymptomatic Chronic Lymphocytic Leukaemia; IgM Monoclonal Gammopathy; Asymptomatic Waldenstrom's Macroglobulinaemia; Immunoglobulin A or G Monoclonal Gammopathy; Smouldering Myeloma; Pre-cancerous; Lymphoproliferative Disorders
MeSH Terms: conditions — Smoldering Multiple Myeloma; Lymphoproliferative Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood Plasma Saliva Bone marrow aspirate
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Cohort 1: Participants with Monoclonal B-Cell Lymphocytosis or Asymptomatic Chronic Lymphocytic Leukaemia
- Cohort 2: Participants with IgM Monoclonal Gammopathy or Asymptomatic Waldenstrom's Macroglobulinaemia
- Cohort 3: Participants with IgA or IgG Monoclonal Gammopathy or Smouldering Myeloma

SUMMARY:
OxPLoreD is an observational cohort study to identify clinical, genomic and immunological predictive markers of progression to malignant disease. Open to individuals diagnosed in the last 3 years with high count MBL, Binet Stage A CLL, Immunoglobulin G/A/M (IgG, IgA, IgM) MGUS, asymptomatic WM not requiring treatment and smouldering myeloma not requiring treatment.

DETAILED DESCRIPTION:
The purpose of the study is to monitor patients with early stage lymphoproliferative disorders not meeting criteria for treatment, including early stage Chronic Lymphocytic Leukaemia (CLL), Monoclonal B-cell Lymphocytosis (MBL), Monoclonal Gammopathy of Uncertain Significance (MGUS), asymptomatic Waldenstroms Macroglobulinaemia (WM) and Smouldering Myeloma (SM).

Each of these disorders has a pre-cancerous phase when abnormalities can be seen in the blood, however treatment may not be required. A minority of people with early stage lymphoproliferative disorders will go on to need treatment for blood or bone marrow cancer.

Currently the investigators do not have a reliable way to predict which of these individuals with these disorders are more likely to develop a blood or bone marrow cancer. By studying a large group of individuals over time we hope to discover more about what factors might predict progression. The investigators may be able to identify markers which identify individuals who are more or less likely to develop blood or bone marrow cancer. These markers might be particular symptoms, gene changes called mutations or levels of particular molecules or cells in the blood or bone marrow. In the longer term this may enable us to identify those people who would benefit from certain types of treatment or from receiving treatment at an earlier stage and also to confidently reassure those who will never progress.

Patients will be studied for up to 5 years with blood, bone marrow and saliva samples taken at key time-points to help answer these questions. In addition to looking for these markers we will also collect information about:

* What it is like to live with one of these conditions
* How many people with these conditions develop other significant medical conditions, such as serious infections, thrombosis (blood clots) or other types of cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed within the previous three years with one of the following:

   1. High count monoclonal B-cell lymphocytosis (MBL) i.e. clonal B-cell population 0.5-4.9 109/L
   2. Rai Stage 0-2/ Binet Stage A or Stage B Chronic Lymphocytic Leukaemia not meeting the IWCLL criteria for treatment
   3. IgG or IgA Monoclonal Gammopathy of Uncertain Significance meeting one of the following criteria:

   i) IgA paraprotein >10g/L or

   ii) IgG paraprotein >15g/L or

   iii) IgA/IgG paraprotein below these cut-offs but kappa:lambda light chain ratio of
   * <0.1 to >3.0 (For OUH participants or sites with no pre-defined cut offs for high risk MGUS) or
   * within the cut off criteria of the local laboratory ranges for high risk MGUS

   iv) Patients not meeting the cut-offs defined in points i) to iii) but who are referred to secondary care e.g. due to general practitioner (GP) concern or for investigation of symptoms

   d. IgM Monoclonal Gammopathy of Uncertain Significance meeting one of the following criteria: i) IgM paraprotein >10g/L or

   ii) IgM paraprotein <10g/L and difference between the kappa and lambda light chains of >50mg/L

   iii) Patients not meeting the cut-offs defined in point i) and ii) but who are referred to secondary care e.g. due to GP concern or investigation of symptoms

   e) Asymptomatic smouldering Waldenstrom's Macroglobulinaemia not meeting the criteria for treatment f) Smouldering myeloma not meeting the criteria for treatment
2. Eastern Cooperative Oncology Group (ECOG) performance status of 0,1 or 2
3. Age 16 years and over
4. Sign written informed consent
5. The patient is willing and able to comply with the protocol for the duration of the study and scheduled follow-up visits and examinations

Exclusion Criteria:

1. Pregnant or breast-feeding women. Pregnant or breast-feeding women may be re-screened following delivery and/or cessation of breastfeeding, as appropriate
2. Previous chemotherapy or immunotherapy for any haematological cancers
3. Treatment with any other investigational agent, or participation in an interventional clinical trial within 28 days prior to enrolment.
4. Patients in cohort 2 or 3 on anticoagulation for a diagnosis of pulmonary embolus or deep vein thrombosis within the last 3 months or with a mechanical heart valve or any other condition causing a significant risk of thromboembolism. Participants who are anticoagulated for atrial fibrillation are eligible, but will be asked to interrupt anticoagulation 3 days prior to bone marrow examination
5. Other psychological, social or medical condition, physical examination finding or laboratory abnormality that the investigator considers would make the patient a poor study candidate or could interfere with protocol compliance or the interpretation of study results.
6. Any other malignancy that requires active surgical or chemotherapeutic Patients on long term hormone therapies (e.g. Tamoxifen) are permitted to enrol at the discretion of investigator, after considering the overall clinical context
7. Any significant concurrent medical resulting in life-expectancy (including but no limited to renal, Hepatic, haematological gastrointestinal, endocrine pulmonary neurological, cerebral or psychiatric disease
8. For cohort 3: Any contraindication for MRI- presence of any metallic foreign body, eGFR <30 and allergy to gadolinium contrast

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study targets three groups of pre-cancerous lymphoproliferative disorders
Sampling Method: Probability Sample
Enrollment: 574 (Actual)
Dates: Start 2019-07-03 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
The identification of predictive markers of progression to malignant disease | Duration of the study (5 years)
  Relevant markers will be identified from the analysis of the clinical data in combination with the genomic and immunological data from the samples collected. The markers will be combined to produce a single probability risk score. The choice of relevant markers will be guided by emerging evidence and techniques under the guidance of the study scientific advisory board.

SECONDARY OUTCOMES:
Patient reported outcome measures (PROM) via approved quality of life questionnaires. | Duration of study (5 years)
  Analysis of approved questionnaires: EORTC CLL17
To study other clinically significant events, not inevitably due to disease progression in this patient cohort | Duration of study (5 years)
  Assessed by analysing suspected unexpected serious adverse reactions (SUSARs) reported
Production of evidence-based standard of care guidelines for the monitoring and follow-up of patients with these pre-cancerous conditions | Duration of study (5 years)
  The identification of relevant markers can be used to create guidelines for optimal monitoring of patients with these pre-cancerous conditions
Patient reported outcome measures (PROM) via approved quality of life questionnaires. | Duration of study (5 years)
  Analysis of approved questionnaires: EORTC NHL-LG20
Patient reported outcome measures (PROM) via approved quality of life questionnaires. | Duration of study (5 years)
  Analysis of approved questionnaires: EORTC QLQ-C30
Patient reported outcome measures (PROM) via approved quality of life questionnaires. | Duration of study (5 years)
  Analysis of approved questionnaires: EORTC QLQ-MY20

CONTACTS AND LOCATIONS:
Overall Officials: Anna Schuh, Principal Investigator — University of Oxford
Locations (17):
- United Kingdom (17):
  - Royal Bournemouth Hospital, Bournemouth
  - Russells Hall Hospital, Dudley
  - James Paget Hospital, Great Yarmouth
  - Leicester Royal Infirmary, Leicester
  - Clatterbridge Cancer Centre, Liverpool
  - Epsom Hospital, London
  - King's College Hospital, London
  - St George's Hospital, London
  - Northern Centre for Cancer Care, Newcastle
  - North Tyneside General Hospital, North Shields
  - Queens Medical Centre, Nottingham
  - Churchill Hospital, Oxford University Hospitals Trust, Oxford
  - Derriford Hospital, Plymouth
  - Poole Hospital, Poole
  - South Tyneside District Hospital, South Shields
  - Sunderland Royal Hospital, Sunderland
  - Musgrove Park Hospital, Taunton

IPD SHARING:
Plan to Share IPD: Undecided